CLINICAL TRIAL: NCT00566397
Title: A Double Blind, Placebo Controlled, Randomized, Multicenter Study Evaluating The Efficacy And Safety Of Eighteen Months Of Treatment With PF 04494700 (TTP488) In Participants With Mild To Moderate Alzheimer's Disease
Brief Title: A Phase 2 Study Evaluating The Efficacy And Safety Of PF 04494700 In Mild To Moderate Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Alzheimer's Disease Cooperative Study (ADCS) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B0341002
Record Dates: First submitted 2007-11-29; First posted 2007-12-03 (Estimated); Last update posted 2018-11-30 (Actual); Status verified 2018-11

CONDITIONS: Alzheimer's Disease
Keywords: RI RI Study Rage Inhibitors
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: PF-04494700
- 2 (Experimental)
  Interventions: Drug: PF-04494700
- 3 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-04494700 — 15 mg for 6 days followed by daily dosing of 5mg
  Arms: 1
Drug: PF-04494700 — 60 mg for 6 days followed by daily dosing of 20mg. Dosing in this arm has been discontinued.
  Arms: 2
Drug: Placebo — Placebo
  Arms: 3

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of PF 04494700 in participants with mild to moderate Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Mini Mental State Exam (MMSE) score between 14-26 (inclusive) at screening.
* Participants must be receiving acetylcholinesterase inhibitors on a stable dose for at least 4 months prior to randomization

Exclusion Criteria:

* Current evidence or history of neurological, psychiatric and any other illness that could contribute to non-Alzheimer's dementia.
* Known history of familial AD or any evidence for early onset AD known or possibly associated with genetic mutations.
* Evidence or history of diabetes mellitus Type 1 or Type 2.
* History or symptoms of autoimmune disorders.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Actual)
Dates: Start 2007-12; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Evaluate the efficacy of PF 04494700 relative to placebo. Change from baseline in a standardized cognitive measure after 18 months of treatment. | 18 Month
Examine the safety and tolerability of PF 04494700 relative to placebo. Adverse events, vital signs, physical exam, neuro exam, 12-lead ECG, lab tests (hematology, blood chemistry, urinalysis) and brain magnetic resonance imaging (MRI). | 18 Month

SECONDARY OUTCOMES:
Evaluate the effects of PF 04494700 on potential biomarkers of RAGE inhibition and amyloid imaging (AV-45, F18 PET) | 18 Month
Evaluate the potential dose response of PF 04494700 | 18 Month
Evaluate the pharmacokinetics and characterize the pharmacokinetic (PK)/ pharmacodynamic (PD) relationship of PF 04494700 to potential biomarkers and relevant efficacy and safety endpoints | 18 Month

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (43):
- United States (43):
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Sun City, Arizona
  - Pfizer Investigational Site, Irvine, California
  - Pfizer Investigational Site, La Jolla, California
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Martinez, California
  - Pfizer Investigational Site, Newport Beach, California
  - Pfizer Investigational Site, Orange, California
  - Pfizer Investigational Site, Palo Alto, California
  - Pfizer Investigational Site, Sacramento, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, San Francisco, California
  - Pfizer Investigational Site, Vista, California
  - Pfizer Investigational Site, New Haven, Connecticut
  - Pfizer Investigational Site, Washington D.C., District of Columbia
  - Pfizer Investigational Site, Jacksonville, Florida
  - Pfizer Investigational Site, Miami Beach, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Ann Arbor, Michigan
  - Pfizer Investigational Site, Grand Rapids, Michigan
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, Beachwood, Ohio
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Pittsburgh, Pennsylvania
  - Pfizer Investigational Site, Providence, Rhode Island
  - Pfizer Investigational Site, Charleston, South Carolina
  - Pfizer Investigational Site, North Charleston, South Carolina
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Salt Lake City, Utah
  - Pfizer Investigational Site, Seattle, Washington
  - Pfizer Investigational Site, Madison, Wisconsin

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0341002&StudyName=A%20Double-Blind%2C%20Placebo-Controlled%2C%20Randomized%2C%20Multicenter%20Study%20Evaluating%20The%20Efficacy%20And%20Safety%20of%20Eighteen%20Months%20Of%20Treatment%20With%20PF-04494700%20%28TTP488%29%20In%20Participants%20With%20Mild%20To%20Moderate%20Alzheimer%27s%20Disease